CLINICAL TRIAL: NCT06087627
Title: Prospective, Non-interventional Observational Study to Characterize Dupilumab Long-term Treatment, Safety and Patient Reported Outcomes in Chronic Nodular Prurigo (Prurigo Nodularis) in Clinical Routine
Brief Title: A Non-interventional Study to Describe the Dupilumab Long-term Treatment, Safety and Patient Reported Outcomes in Chronic Nodular Prurigo (Prurigo Nodularis) in Clinical Routine
Acronym: CLEAR PN
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17933; U1111-1290-5823 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PN treatment: Participants ≥ 18 years suffering from moderate-to-severe PN who receive long-term dupilumab treatment for PN in a real-world setting in Germany.
  Interventions: Drug: Dupilumab SAR231893 (REGN668)

INTERVENTIONS:
Drug: Dupilumab SAR231893 (REGN668) — Subcutaneous injection, standard of care as prescribed by treating physician (no investigational drug provided)
  Other Names: Dupixent®

SUMMARY:
Prurigo nodularis (PN) is a skin disease characterized by the presence of single to multiple symmetrically distributed, intensively itching nodules. The main symptom is uncontrollable itching leading to prolonged, repetitive, and uncontrollable rubbing, scratching which in turn causes injuries to the skin. In recent years, number of studies evaluating PN, the affected population and the disease burden has increased but PN remains still understudied. This non-interventional study is intended to describe the long-term effectiveness of dupilumab (Dupixent®) in participants aged 18 years or older and suffering from moderate-to-severe PN who receive dupilumab for PN treatment in a real-world setting in Germany according to the prescribing information (Summary of Product Characteristics [SmPC]). The decision to initiate dupilumab treatment is made by the treating physician and participant according to the participant's medical need and to the standard of best medical practice. This decision is made independently and before data inclusion in this non-interventional study.

DETAILED DESCRIPTION:
The individual observational period is planned to be up to 2 years, with assessments at baseline, one month after baseline and afterwards, every 3 months in the 1st and every 6 months in the 2nd year after dupilumab initiation, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years of age at baseline visit
* Signed written informed consent
* New initiation with dupilumab or in whom treatment with dupilumab was started within the last 7 days for moderate to severe prurigo nodularis according to the prescribing information/Summary of Product Characteristics (SmPC)
* Patients who received the initial diagnosis of PN

Exclusion Criteria:

* Patients who have a contraindication to dupilumab according to the current prescribing information label/SmPC
* Patients who have been treated for more than 7 days with dupilumab
* Any acute or chronic condition that, in the treating physician´s opinion, would limit the patient´s ability to complete questionnaires or to participate in this study or impact the interpretation of the results
* Participation in an ongoing interventional or observational study that might, in the treating physician´s opinion, influence the assessments for the current study

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants ≥ 18 years suffering from moderate-to-severe PN who receive long-term dupilumab treatment for PN in a real-world setting in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of participants with Investigator Global Assessment Prurigo Nodularis Stage (IGA-CPG-S) score 0 or 1 in Month 6 | Month 6
  IGA CPG-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe prurigo nodularis (PN).
Percentage (%) of participants with greater than or equal to (≥) 4-point improvement (reduction) in Worst Itch Numerical Rating Scale (WI-NRS) from baseline to Month 6 | Baseline, Month 6
  WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity.

SECONDARY OUTCOMES:
Characterization of the participants who receive dupilumab for PN: Socio-demographic data | Baseline
Characterization of the participants who receive dupilumab for PN: Medical history of disease | Baseline
Characterization of the participants who receive dupilumab for PN: Previous PN treatment (including balneophototherapy and/or UV therapy) | Baseline
Characterization of the participants who receive dupilumab for PN: Current PN treatment (INN, topical and/or systemic) | Baseline, Months 1, 3, 6, 9, 12, 18 and 24
Characterization of the participants who receive dupilumab for PN: Concomitant medication (INN) | Baseline, Months 1, 3, 6, 12 and 24
Characterization of the participants who receive dupilumab for PN: Presence of relevant comorbidities or of other prurigo subtypes | Baseline
  Relevant comorbidities include presence of associated atopic comorbidities or type 2 inflammatory diseases.
Characterization of the participants who receive dupilumab for PN: Biomarker levels (if available) | Baseline
Characterization of the participants who receive dupilumab for PN: Laboratory results (if available) | Baseline
  Data for any of the following laboratory parameters will be collected as available in routine clinical practice and expressed in the units relevant for the respective parameter: bilirubin, aspartate amino transferase (AST), alanine amino transferase (ALT), gamma glutamyl transferase (gamma GT), alkaline phosphatase, differential blood count, ferritin, erythrocyte sedimentation rate, C-reactive protein.
Characterization of the participants who receive dupilumab for PN: Reasons for initiation of dupilumab treatment | Baseline
Effectiveness of dupilumab: Patient Global Impression of Change (PGIC) of PN disease at month 1, month 3, month 6, month 12, and month 24 of dupilumab therapy | Months 1, 3, 6, 12 and 24
  PGIC is a 7-point scale to assess patient health and determine if there has been an improvement or decline in clinical status. Patients are asked to rate their overall status since the start of the study from "very much improved" to "very much worse". Scores range from 1 to 7, with higher score indicating worse health status.
Effectiveness of dupilumab: Change in Prurigo Control Test (PCT) from baseline to month 6, month 12, and month 24 after initiation of dupilumab therapy | Baseline to Months 6, 12 and 24
  PCT is a self-administered, simple 5-item tool. A score between 0 and 4 is assigned to every answer option. Subsequently, the scores for all 5 questions are summed up. Accordingly, the minimum and maximum PCT scores are 0 and 20, with higher scores indicating a higher level of disease control.
Effectiveness of dupilumab: Change in Dermatology Life Quality Index (DLQI) from baseline to month 3, month 6, month 9, month 12, month 18, and month 24 after initiation of dupilumab therapy | Baseline to Months 3, 6, 9, 12, 18 and 24
  DLQI is developed to measure dermatology specific Health-Related Quality of Life (HRQoL) in adult participants. It comprises of set of 10 questions assessing the impact of skin disease on participants' HRQoL over the previous week. Responses to each question were assessed on a 4-point Likert scale ranged from 0 (not at all) to 3 (very much). Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Effectiveness of dupilumab: Change in Sleep Numerical Rating Scale (Sleep-NRS) from baseline to month 6, month 9, month 12, month 18, and month 24 after initiation of dupilumab therapy | Baseline to Months 6, 9, 12, 18 and 24
  Sleep-NRS was used to measure sleep intensity. Participants were asked to rate their sleep quality on their past night upon awakening, using a 11-point NRS ranging from 0 to 10, where 0 = worst possible sleep and 10 = best possible sleep. Higher scores indicated less severity.
Effectiveness of dupilumab: Percentage (%) of participants with ≥ 4-point improvement (reduction) in WI-NRS from baseline to month 1, month 3, month 9, month 12, month 18, and month 24 after initiation of dupilumab therapy | Baseline to Months 1, 3, 9, 12, 18 and 24
  WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity.
Effectiveness of dupilumab: Percentage (%) of participants with IGA-CPG activity (IGA-CPG-A) score of 0 or 1 at month 1, month 3, month 6, month 9, month 12, month 18, and month 24 after initiation of dupilumab therapy | Months 1, 3, 6, 9, 12, 18 and 24
  The IGA CPG-A is an instrument used to assess the overall activity of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4: where 0 = clear (0% nodules showing excoriations/crusts), 1 = almost clear (up to 10% nodules showing excoriations/crusts), 2 = mild (11-25% nodules showing excoriations/crusts), 3 = moderate (26-75% nodules showing excoriations/crusts) and 4 = severe (76-100% of nodules showing excoriations/crusts). Higher scores indicate severe PN.
Effectiveness of dupilumab: Percentage (%) of participants with IGA-CPG-S score of 0 or 1 in month 1, month 3, month 9, month 12, month 18, and month 24 after initiation of dupilumab therapy | Months 1, 3, 9, 12, 18 and 24
  IGA CPG-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe PN.
Effectiveness of dupilumab: Percentage (%) of participants with Patient Benefit Index-Pruritus (PBI-P) ≥ 1 at month 6, month 12, and month 24 of dupilumab therapy | Months 6, 12 and 24
  PBI-P is a validated questionnaire where, prior to treatment, individual participants determine how different benefits of therapy would be relevant for them. After treatment, participants will be asked to evaluate the extent to which the benefits they indicated were important to them were, in fact, realized. From all the items taken together, a weighted total benefit value is calculated, which represents the patient relevant therapy benefits. The mean score greater than 1 is considered to represent a clinically relevant improvement. The items are rated on a 5-point scale with values from 0 (not at all) to 4 (very), allowing for 'does/did not apply to me' = 5; and missing value = -9. Higher scores indicate better outcome.
Effectiveness of dupilumab: Change in Hospital Depression and Anxiety Score (HADS total score) from baseline to month 6, month 12, and month 24 of dupilumab therapy | Baseline to Months 6, 12 and 24
  HADS is a 14-item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale comprised of 7 items with a scoring range from 0 (less severity of anxiety and depression) to 21 (greater severity of anxiety and depression symptoms) for each subscale. The total HADS score ranges from 0 (less severity) to 42 (more severity), with a high score indicative of severe anxiety and/or depression level.
Effectiveness of dupilumab: Percentage of participants who achieve ≥ 75% healed lesions from Prurigo Activity Score (PAS) from baseline to month 3, month 6, month 12, and month 24 of dupilumab therapy | Baseline to Months 3, 6, 12 and 24
  The items of the PAS evaluate the type (visible lesions: item 1a; predominant lesions: item1b), estimated number (item 2), distribution (item 3, 4) and size (biggest lesion: item 6a; representative lesion: item 6b) of pruriginous lesions, the representative body area and exact number of lesions (item 5), the activity in terms of percentage of pruriginous lesions with excoriations/crusts on top (reflecting active scratching; item 7a) and the percentage of healed pruriginous lesions (reflecting healing of CPG; item 7b).
Effectiveness of dupilumab: Number of sick-leave days at work due to PN during the last 12 months before baseline and since the last visit after starting dupilumab treatment | Baseline, Month 1, 3, 6, 12 and 24
Effectiveness of dupilumab: Number and duration of hospitalization due to PN during the last 12 months after 12 and 24 months of dupilumab therapy | Baseline to Month 12 and Month 24
Pharmacodynamics of dupilumab: Pharmacodynamic response for selected biomarkers (total IgE, blood eosinophils) at month 12 and month 24 after initiation of dupilumab therapy | Month 12, Month 24
Treatment patterns during real-world use of dupilumab: Dupilumab dose regimens used over the study, and the duration with each regimen | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Percentage of participants whose dose (either the frequency or the strength) increased from starting regimen and reasons | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Percentage of participants whose dose (either the frequency or the strength) decreased from the starting regimen and reasons | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Percentage of participants discontinuing dupilumab, including temporary or permanent discontinuation | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Type of treatment switched to after discontinuing dupilumab | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Duration of use, drug survival of dupilumab | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Number of gaps in dupilumab treatment and longest gap length | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Concomitant therapies taken for PN | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Reason for switching or discontinuing dupilumab | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Time from baseline to self-administer dupilumab at home | Baseline to Month 24
Safety: Occurrence and type of Treatment-Emergent Adverse Events (TEAEs) during the observational period | Baseline to Month 24
Safety: Occurrence and type of dupilumab-related TEAEs during the observational period | Baseline to Month 24
Safety: Event rate (per patient year) by type of TEAEs during the observational period | Baseline to Month 24
Safety: Event rate (per patient year) by type of dupilumab-related TEAEs during the observational period | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Number of gaps in dupilumab treatment | Baseline to Month 24
Treatment patterns during real-world use of dupilumab: Longest gap length in dupilumab treatment | Baseline to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Germany (11):
  - Investigational Site Number: 013, Adernach
  - Investigational site number: 001, Berlin
  - Investigational Site Number: 002, Berlin
  - Investigational Site Number: 023, Chemnitz
  - Investigational Site Number: 005, Düren
  - Investigational Site Number: 004, Düsseldorf
  - Investigational Site Number: 007, Hamburg
  - Investigational Site Number: 016, Leipzig
  - Investigational Site Number: 031, Mainz
  - Investigational Site Number: 022, Potsdam
  - Investigational Site Number: 024, Potsdam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org